CLINICAL TRIAL: NCT02649465
Title: Pleiotropic Effects and Safety of Sodium Glucose Co-transporter 2 Inhibitor Versus Sulfonylurea in Patients With Type 2 Diabetes and Non-alcoholic Fatty Liver
Brief Title: SGLT2 Inhibitor Versus Sulfonylurea on Type 2 Diabetes With NAFLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kanazawa University (Other)
Collaborators: Kowa Company, Ltd. (Industry)
Responsible Party: Principal Investigator, Toshinari Takamura, MD, PhD, Department of Disease Control and Homeostasis, Kanazawa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRB4180005
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SGLT2 inhibitor (Active Comparator): N=20 SGLT2 inhibitor dosage (Tofogliflozin): a dose of 20mg once daily for 48 weeks.
  Interventions: Drug: Tofogliflozin
- Sulfonylurea (Active Comparator): N=20 Sulfonylurea (Glimepiride): an initial dose of 0.5 mg once daily for 48 weeks.
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Tofogliflozin — The group receiving Tofogliflozin (at a dose of 20mg once daily) for 48 weeks
  Other Names: DEBERZA
  Arms: SGLT2 inhibitor
Drug: Glimepiride — Sulfonylurea dosage (Glimepiride): dosing from 0.5 mg for initial 4 weeks. Then, if there is no adverse effect or no improvement of glucose metabolism, glimepiride is escalated to 6 mg once daily.
  Arms: Sulfonylurea

SUMMARY:
The clinicopathological analyses revealed that reduction in HbA1c and use of insulin independently contribute to the reduction in liver fibrosis scores during the histological course of NAFLD development. These findings led us to hypothesize that glycemic control and insulin ameliorate or protect against the histological progression of liver fibrosis in patients with NAFLD.

In the present study, we investigated the efficacy of SGLT2 inhibitor tofogliflozin and sulfonylurea glimepiride, which lower glucose levels similarly with reduction and elevation in circulating insulin levels, respectively, in NAFLD patients with type 2 diabetes for 48 weeks by examining liver histology, as well as hepatic enzymes, metabolic markers, and hepatic gene expression profiles.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD), ranging from simple fatty liver to nonalcoholic steatohepatitis (NASH), is a liver phenotype of metabolic disorders, such as diabetes, obesity, and metabolic syndrome. NAFLD and type 2 diabetes share epidemiological and pathophysiological features. Specifically, hyperglycemia is closely associated with liver fibrosis, which is associated with liver cirrhosis, hepatocellular carcinoma, and prognosis in patients with NASH.

To date, some anti-diabetic agents have been tested in patients with NAFLD. The guidelines in the Asian Pacific, European, and American association recommended the administration of PPAR gamma agonist (pioglitazone) and glucagon-like peptide receptor agonists (GLP1RA) for the treatment of diabetes with NAFLD/NASH. However, there are concerns about adverse effects such as weight gain, edema, fractures, and carcinogenesis in pioglitazone or gastrointestinal adverse effects and medication burden as an injection in GLP1 RA. In addition, because all of these anti-diabetic agents significantly reduced glycemic levels compared with placebo, liver histological improvement may be theoretically attributable to glucose reduction itself.

Both sodium-glucose cotransporter 2 (SGLT2) inhibitors and sulfonylureas are chosen as the second-line therapy when glycemic control cannot be achieved with metformin or as the first-line therapy when metformin is contraindicated or not tolerated. In animal models of NAFLD/NASH, SGLT2 inhibitors protect against steatosis, inflammation, and fibrosis. Previous clinical trials have demonstrated that SGLT2 inhibitors exert protective effects on liver enzymes and liver steatosis in patients with NAFLD/NASH. However, these studies lack a control group or histological examination, which precludes meaningful conclusions since the natural course of the disease or tight glycemic control may ameliorate liver histology in some patients with NAFLD. Sulfonylureas are still reliable and potent antidiabetic agents in insulinopenic patients with type 2 diabetes and therefore are used as the second-line therapy, especially when the cost is a significant issue. Besides, sulfonylureas reduce glucose and elevate weight, which may render positive and negative effects, respectively, on liver pathology in NAFLD/NASH. In the phase 3 trial, canagliflozin was non-inferior to glimepiride for reduction of HbA1c at 52 weeks. However, the differences between SGLT2 inhibitors and sulfonylureas on NAFLD patients with type 2 diabetes under similar glucose reduction remain uncertain.

ELIGIBILITY:
The trial entry criteria are based on:

1. A diagnosis of "definite" NAFLD on liver biopsy obtained within 3 months of screening.
2. ≥20 years of age at the time of the initial screening.
3. Patients with type 2 diabetes mellitus at the time of screening need to have glycemic control (HbA1c of ≥7%) and have been managed by either diet and/or a stable dose of hypoglycemic agents for at least 4 weeks.

Exclusion Criteria

1. Hepatic virus infections (hepatitis B and C, cytomegalovirus, and Epstein-Barr virus), autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, hemochromatosis, alpha 1-antitrypsin deficiency, Wilson's disease, history of parenteral nutrition.
2. Use of agents known to induce steatosis (e.g., valproate, amiodarone, or vitamin E)
3. Hepatic injury caused by substance abuse.
4. Current consumption of more than 20 g of alcohol daily.
5. Hepatic decompensation, such as hepatic encephalopathy, ascites, variceal bleeding
6. Elevated serum bilirubin level of more than two-fold the upper normal limit.
7. Tofogliflozin or glimepiride hypersensitivity or contraindications.
8. History of type 1 diabetes.
9. History of ketoacidosis.
10. History of symptoms of severe hypoglycemia.
11. Treatment with SGLT2 inhibitor including tofogliflozin within 4 weeks of screening.
12. Treatment with glinide and sulfonylurea use within 4 weeks of screening.
13. Concomitant corticosteroid therapy uses within 4 weeks of screening.
14. Poorly controlled unstable diabetes (ketoacidosis or an increase in HbA1c of >3% in the 12 weeks before screening).
15. Poorly controlled hypertension or systolic blood pressure of >160 mmHg or diastolic blood pressure of >100 mmHg.
16. Artificial dialysis or moderate renal dysfunction.
17. Poorly controlled dyslipidemia.
18. Presence of a severe health problem, not being suitable for the study.
19. Pregnant or breastfeeding.
20. Inability to participate in the study (including psychiatric and psychosocial problems), as assessed by the investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The improvement in histologic features of NAFLD | 48 weeks

SECONDARY OUTCOMES:
Change from baseline in liver enzymes | 48 weeks
Change from baseline in body composition | 48 weeks
Change from baseline in fasting plasma glucose level and glucose metabolism assessed with arginine tolerance test | 48 weeks
Changes from baseline in organ-specific insulin sensitivity and glucagon response during a euglycemic hyperinsulinemic clamp study | 48 weeks
Change from baseline in lipid profile | 48 weeks
Change from baseline in renal function and electrolyte balances | 48 weeks
Change from baseline in oxidative stress | 48 weeks
Change from baseline in cytokine (TNF-alpha, leptin, adiponectin) levels | 48 weeks
Change from baseline in hepatokine (Selenoprotein P, LECT2) levels | 48 weeks
Change from baseline in organ-specific fat accumulation | 48 weeks
Change from baseline in oxidative and non-oxidative glucose disposal | 48 weeks
Change from baseline in respiratory quotients | 48 weeks
Change from baseline in energy expenditure | 48 weeks
Change from baseline in autonomic nerve function. | 48 weeks
Changes from baseline in minerals and bone metabolism | 48 weeks
Changes from baseline in endothelial functions | 48 weeks
Changes from baseline in fatty acids profiles | 48 weeks
Factors associated with the changes in autonomic nerve function, organ-specific fat accumulation, and glucagon response. | 48 weeks
Changes from baseline in gene expression profiles in the liver and blood cells | 48 weeks
Changes from baseline in microRNAs and exosome contents | 48 weeks
Epigenomic changes from baseline in genes of the liver and blood cells | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshinari Takamura, MD,PhD, Study Chair — Department of Endocrinology and Metabolism, Kanazawa University Graduate School of Medical Sciences,
Locations (1):
- Kanazawa University Graduate School of Medical Sciences, Kanazawa, Ishikawa-ken, Japan

IPD SHARING:
Plan to Share IPD: No
The datasets are not readily available because several studies are ongoing using the datasets in the present study. Requests to access the datasets should be directed to the correspondence author. We will open raw data with the appropriate institutional ethics committee's prior approval.

REFERENCES:
- [Derived] Takeshita Y, Honda M, Harada K, Kita Y, Takata N, Tsujiguchi H, Tanaka T, Goto H, Nakano Y, Iida N, Arai K, Yamashita T, Mizukoshi E, Nakamura H, Kaneko S, Takamura T. Comparison of Tofogliflozin and Glimepiride Effects on Nonalcoholic Fatty Liver Disease in Participants With Type 2 Diabetes: A Randomized, 48-Week, Open-Label, Active-Controlled Trial. Diabetes Care. 2022 Sep 1;45(9):2064-2075. doi: 10.2337/dc21-2049. PMID 35894933
- [Derived] Takeshita Y, Kanamori T, Tanaka T, Kaikoi Y, Kita Y, Takata N, Iida N, Arai K, Yamashita T, Harada K, Gabata T, Nakamura H, Kaneko S, Takamura T. Study Protocol for Pleiotropic Effects and Safety of Sodium-Glucose Cotransporter 2 Inhibitor Versus Sulfonylurea in Patients with Type 2 Diabetes and Nonalcoholic Fatty Liver Disease. Diabetes Ther. 2020 Feb;11(2):549-560. doi: 10.1007/s13300-020-00762-9. Epub 2020 Jan 20. PMID 31956961